CLINICAL TRIAL: NCT05558410
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Suzetrigine for Acute Pain After an Abdominoplasty
Brief Title: Evaluation of Efficacy and Safety of Suzetrigine for Acute Pain After an Abdominoplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX22-548-105
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo matched to Suzetrigine (SUZ) and Hydrocodone bitartrate/acetaminophen (HB/APAP) for 48 hours.
  Interventions: Drug: Placebo (matched to SUZ); Drug: Placebo (matched to HB/APAP)
- Hydrocodone bitartrate/acetaminophen (HB/APAP) (Active Comparator): Participants received HB 5 milligrams (mg)/ APAP 325 mg every 6 hours (q6h) for 48 hours.
  Interventions: Drug: HB/APAP; Drug: Placebo (matched to SUZ)
- Suzetrigine (SUZ) (Experimental): Participants received SUZ [100 mg as first dose, followed by 50 mg every 12 hours (q12h)] for 48 hours.
  Interventions: Drug: Suzetrigine (SUZ); Drug: Placebo (matched to HB/APAP)

INTERVENTIONS:
Drug: Suzetrigine (SUZ) — Tablets for oral administration.
  Other Names: VX-548
  Arms: Suzetrigine (SUZ)
Drug: HB/APAP — Capsules for oral administration.
  Arms: Hydrocodone bitartrate/acetaminophen (HB/APAP)
Drug: Placebo (matched to SUZ) — Placebo matched to SUZ for oral administration.
  Arms: Hydrocodone bitartrate/acetaminophen (HB/APAP); Placebo
Drug: Placebo (matched to HB/APAP) — Placebo matched to HB/APAP for oral administration.
  Arms: Placebo; Suzetrigine (SUZ)

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of Suzetrigine (SUZ) in treating acute pain after an abdominoplasty.

ELIGIBILITY:
Key Inclusion Criteria:

* Before Surgery

  * Participant scheduled to undergo a standard ("full") abdominoplasty procedure
* After Surgery

  * Participant is lucid and able to follow commands and able to swallow oral medications
  * All analgesic guidelines were followed during and after the abdominoplasty
  * Abdominoplasty procedure duration less than or equal to (≤3) hours

Key Exclusion Criteria:

* Before Surgery

  * Prior history of abdominoplasty
  * History of Intra-abdominal and/or pelvic surgery that resulted into complications
  * History of cardiac dysrhythmias within the last 2 years requiring anti-arrhythmia treatment(s)
  * Any prior surgery within 1 month before the first study drug dose
* After Surgery

  * Participant had a non standard abdominoplasty, collateral procedures during the abdominoplasty or any surgical complications during the abdominoplasty
  * Participant had a medical complication during the abdominoplasty that, in the opinion of the investigator, should preclude randomization

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1118 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-09-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Shoals Medical Trials Inc., Sheffield, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Alliance Research Institute, LLC, Canoga Park, California
  - New Hope Research Development, Tarzana, California
  - Atlanta Center for Medical Research | Atlanta, GA, Atlanta, Georgia
  - Kansas Spine and Specialty Hospital, Wichita, Kansas
  - HD Research LLC | First Surgical Hospital, Bellaire, Texas
  - HD Research LLC | Houston Heights Hospital, Houston, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - South Texas Spine & Surgical Hospital, San Antonio, Texas
  - JBR Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Hydrocodone Bitartrate/Acetaminophen (HB/APAP) | Suzetrigine (SUZ)
Started | 223 | 448 | 447
Safety Set (Safety set included all participants who received at least 1 dose of study drug.) | 222 (Due to an error in dispensing study drug kits at 1 site, 1 participant who was randomized to placebo group received 1 dose of active SUZ. Therefore, the participant was counted in the placebo group for the full analysis set (FAS) and in the SUZ group for the Safety Set.) | 448 | 448 (Due to an error in dispensing study drug kits at 1 site, 1 participant who was randomized to placebo group received 1 dose of active SUZ. Therefore, the participant was counted in the placebo group for the full analysis set (FAS) and in the SUZ group for the Safety Set.)
Completed | 206 | 426 | 423
Not Completed | 17 | 22 | 24
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Withdrawal of consent (not due to AE) | 3 | 2 | 2
Not completed — Lost to Follow-up | 10 | 17 | 19
Not completed — Death | 1 | 0 | 0
Not completed — Other non-compliance | 0 | 1 | 2
Not completed — Sponsor Decision | 1 | 0 | 0
Not completed — Other | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of the study drug.
Groups:
- Placebo: Participants received placebo matched to SUZ and HB/APAP for 48 hours.
- Hydrocodone Bitartrate/Acetaminophen (HB/APAP): Participants received HB 5 mg/ APAP 325 mg q6h for 48 hours.
- Suzetrigine (SUZ): Participants received SUZ (100 mg as first dose, followed by 50 mg q12h) for 48 hours.
- Total: Total of all reporting groups
Arm/Group | Placebo | Hydrocodone Bitartrate/Acetaminophen (HB/APAP) | Suzetrigine (SUZ) | Total
Number analyzed (Participants) | 223 | 448 | 447 | 1118
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (8.5) | 42.1 (8.7) | 41.5 (9.1) | 41.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220 | 441 | 437 | 1098
  Male | 3 | 7 | 10 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 73 | 157 | 150 | 380
  Not Hispanic or Latino | 150 | 288 | 297 | 735
  Missing | 0 | 3 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 155 | 316 | 307 | 778
  Black or African American | 62 | 114 | 123 | 299
  Asian | 0 | 9 | 7 | 16
  American Indian or Alaska Native | 1 | 0 | 5 | 6
  Native Hawaiian or other Pacific Islander | 1 | 5 | 3 | 9
  Other | 2 | 0 | 0 | 2
  Multiracial | 2 | 4 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of the Pain Intensity Difference (SPID) as Recorded on a Numeric Pain Rating Scale (NPRS) From 0 to 48 Hours (SPID48) SUZ Compared to Placebo
Description: SPID was calculated as the sum of the product of time (in hours) elapsed since previous measurements and pain intensity difference. Pain intensity difference was calculated by subtracting the baseline pain intensity score from the pain intensity score at each postdose time point (using pain rating score range: 0 =no pain to 10 =worst possible pain). SPID48 was calculated from 0 to 48 hours and the score range was -480 (worst score) to 480 (best score).
Time Frame: 0 to 48 hours After First Dose of Study Drug
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 223 | 447
units on a scale | 70.1 (6.1) | 118.4 (4.3)
Statistical Analysis 1: Comparison: Placebo vs Suzetrigine (SUZ); Test type: Superiority; p < 0.0001, ANCOVA

2. Secondary Outcome: Time-weighted Sum of the Pain Intensity Difference (SPID) as Recorded on a Numeric Pain Rating Scale (NPRS) From 0 to 48 Hours (SPID48) SUZ Compared to HB/APAP
Description: SPID was calculated as the sum of the product of time (in hours) elapsed since previous measurements and pain intensity difference. Pain intensity difference was calculated by subtracting the baseline pain intensity score from the pain intensity score at each post dose time point (using pain rating score range: 0 =no pain to 10 =worst possible pain). SPID48 was calculated from 0 to 48 hours and the score range was -480 (worst score) to 480 (best score).
Time Frame: 0 to 48 hours After First Dose of Study Drug
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Hydrocodone Bitartrate/Acetaminophen (HB/APAP) | Suzetrigine (SUZ)
Number analyzed (Participants) | 448 | 447
units on a scale | 111.8 (4.3) | 118.4 (4.3)
Statistical Analysis 1: Comparison: Hydrocodone Bitartrate/Acetaminophen (HB/APAP) vs Suzetrigine (SUZ); Test type: Superiority; p = 0.2781, ANCOVA

3. Secondary Outcome: Time to Greater Than or Equal to (≥) 2-point Reduction in NPRS, SUZ Compared to Placebo
Description: Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain.
  The time to ≥2-point reduction in NPRS from baseline was the time elapsed from the first dose of study drug until the first time the participant had at least a 2-point reduction in NPRS scores from baseline. Participants who did not reach at least a 2-point reduction in NPRS from baseline by 48 hours were censored at 48 hours.
Time Frame: From Baseline Up to 48 Hours After First Dose of Study Drug
Population: FAS.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 223 | 447
minutes | 480 [477 to 705] | 119 [90 to 180]
Statistical Analysis 1: Comparison: Placebo vs Suzetrigine (SUZ); Test type: Superiority; p < 0.0001, Log Rank

4. Secondary Outcome: Time to ≥1-point Reduction in NPRS, SUZ Compared to Placebo
Description: Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain.
  The time to ≥1-point reduction in NPRS from baseline was the time elapsed from the first dose of study drug until the first time the participant had at least a 1-point reduction in NPRS scores from baseline. Participants who did not reach at least a 1-point reduction in NPRS from baseline by 48 hours were censored at 48 hours.
Time Frame: From Baseline Up to 48 Hours After First Dose of Study Drug
Population: FAS.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 223 | 447
minutes | 91 [60 to 180] | 34 [32 to 55]
Statistical Analysis 1: Comparison: Placebo vs Suzetrigine (SUZ); Test type: Superiority; p < 0.0001, Log Rank

5. Secondary Outcome: Percentage of Participants Reporting Good or Excellent on the Patient Global Assessment (PGA) Scale, SUZ Compared to Placebo
Description: The PGA is a single-item assessment of patient perceptions of the method of pain control with the study drug and is evaluated on a 4-point Likert scale as: (poor, fair, good, or excellent). Percentage of participants who reported good or excellent on the PGA scale were reported. Participants who discontinued study drug or had missing PGA at 48 hours were considered to not have reported good or excellent on the PGA.
Time Frame: At 48 hours
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 223 | 447
percentage of participants | 49.8 | 67.8
Statistical Analysis 1: Comparison: Placebo vs Suzetrigine (SUZ); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

6. Secondary Outcome: Incidence of Vomiting or Nausea, SUZ Compared to HB/APAP
Description: The incidence with the events of vomiting or nausea during the specified time frame was reported.
Time Frame: From Baseline Up to Day 19
Population: Safety set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Hydrocodone Bitartrate/Acetaminophen (HB/APAP) | Suzetrigine (SUZ)
Number analyzed (Participants) | 448 | 448
percentage of participants | 33.5 | 20.3
Statistical Analysis 1: Comparison: Hydrocodone Bitartrate/Acetaminophen (HB/APAP) vs Suzetrigine (SUZ); Test type: Superiority; p < 0.0001, Pearson's chi-squared test

7. Secondary Outcome: Time-weighted SPID as Recorded on the NPRS From 0 to 24 Hours (SPID24), SUZ Compared to Placebo
Description: SPID was calculated as the sum of the product of time (in hours) elapsed since previous measurements and pain intensity difference. Pain intensity difference (PID) was calculated by subtracting the baseline pain intensity score from the pain intensity score at each post dose time point (NPRS range: 0 = no pain to 10 = worst possible pain). Time-weighted SPID was calculated as the sum of the PIDs at each post-dose time point multiplied by the time interval (in hours) between each time point. SPID 24 was calculated from 0 to 24 hours and the score range was -240 (worst score) to 240 (best score).
Time Frame: 0 to 24 Hours After First Dose of Study Drug
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 223 | 447
units on a scale | 24.2 (2.8) | 48.0 (2.0)
Statistical Analysis 1: Comparison: Placebo vs Suzetrigine (SUZ); Test type: Superiority; p < 0.0001, ANCOVA

8. Secondary Outcome: Time to First Use of Rescue Medication, SUZ Compared to Placebo
Description: Time to first use of rescue medication is the time from the first dose of study drug until the first use of rescue medication. Participants who did not take any rescue medication within 48 hours were censored at 48 hours.
Time Frame: 0 to 48 Hours After First Dose of Study Drug
Population: FAS.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 223 | 447
minutes | 115 [100 to 132] | 186 [158 to 212]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.0001, Log Rank

9. Secondary Outcome: Percentage of Participants Using Rescue Medication From 0 to 48 Hours, SUZ Compared to Placebo
Time Frame: 0 to 48 Hours After First Dose of Study Drug
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 223 | 447
percentage of participants | 87.9 | 81.0
Statistical Analysis 1: Comparison: Placebo vs Suzetrigine (SUZ); Test type: Superiority; p = 0.0237, Cochran-Mantel-Haenszel

10. Secondary Outcome: Total Rescue Medication Usage, SUZ Compared to Placebo
Time Frame: 0 to 48 Hours After First Dose of Study Drug
Population: FAS.
Measure: Median (Full Range); unit: milligram
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 223 | 447
milligram | 1200 [0 to 3200] | 800 [0 to 3200]
Statistical Analysis 1: Comparison: Placebo vs Suzetrigine (SUZ); Test type: Superiority; p = 0.0080, Wilcoxon rank-sum

11. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Day 19
Population: Safety set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Hydrocodone Bitartrate/Acetaminophen (HB/APAP) | Suzetrigine (SUZ)
Number analyzed (Participants) | 222 | 448 | 448
Participants
  Participants with TEAEs | 125 | 272 | 224
  Participants with SAEs | 5 | 7 | 11

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 19
Groups:
- HB/APAP: Participants received HB 5 mg/ APAP 325 mg q6h for 48 hours.
Arm/Group | Placebo | HB/APAP | Suzetrigine (SUZ)
All-Cause Mortality (participants affected / at risk) | 1/222 | 0/448 | 0/448
Serious Adverse Events (participants affected / at risk) | 5/222 | 7/448 | 11/448
Other Adverse Events (participants affected / at risk) | 94/222 | 201/448 | 146/448
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=222) | HB/APAP (N=448) | Suzetrigine (SUZ) (N=448)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Infected seroma (Infections and infestations) | 0 | 0 | 1
Medical device site infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 2 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 1 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=222) | HB/APAP (N=448) | Suzetrigine (SUZ) (N=448)
Constipation (Gastrointestinal disorders) | 24 | 39 | 47
Nausea (Gastrointestinal disorders) | 56 | 147 | 85
Dizziness (Nervous system disorders) | 17 | 24 | 18
Headache (Nervous system disorders) | 11 | 32 | 19
Hypotension (Vascular disorders) | 15 | 16 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT05558410/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT05558410/SAP_001.pdf